CLINICAL TRIAL: NCT02205840
Title: A Multicenter, Randomized, Double-masked and Placebo-controlled Study Evaluating the Efficacy and Safety of SI-614 Ophthalmic Solution in Patients With Dry Eye
Brief Title: A Clinical Study Evaluating the Safety and Efficacy of SI-614 Ophthalmic Solution in Patients With Dry Eye.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seikagaku Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 614/1131
Record Dates: First submitted 2014-07-30; First posted 2014-07-31 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SI-614 (Experimental)
  Interventions: Drug: SI-614
- Placebo Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: SI-614 — 1 drop in each eye
  Arms: SI-614
Drug: Vehicle — 1 drop in each eye
  Arms: Placebo Vehicle

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of SI-614 solution compared with placebo solution in treating patients with dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Have provided written informed consent
* Have dry eye in both eyes

Exclusion Criteria:

* Use of contact lenses
* Have an uncontrolled systemic disease
* Have an uncontrolled psychiatric condition, or substance or alcohol abuse
* Women who is pregnant, nursing or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Corneal staining score | Up to 28 days
Symptom score | Up to 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Andover, Massachusetts, United States